CLINICAL TRIAL: NCT07272668
Title: Metabolic Availability of Tryptophan in Cornmeal in Healthy Adults >60 Yrs
Brief Title: MA of Tryptophan in Cornmeal in Healthy Adults>60y
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Associate Scientist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3568
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: Protein Absorption and Amino Acid Availability
Keywords: elderly; healthy; tryptophan; amino acid availability; metabolic availability; indicator amino acid oxidation; iaao; stable isotopes
MeSH Terms: interventions — Tryptophan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MA of tryptophan in maize (Experimental): Apply the IAAO method to determine the metabolic availability of tryptophan in maize prepared by moist cooking method
  Interventions: Other: Tryptophan

INTERVENTIONS:
Other: Tryptophan — 4 different tryptophan test levels 0.5, 1, 1.5 and 2 mg.kg-1.day.1
  Other Names: maize

SUMMARY:
The world's population will reach 12 billion by this century's end. As the human population increases, the world faces the continuous challenge of optimizing a limited food supply. Protein is the key determinant of growth and bodily function. Recently, our group showed that current protein recommendations for adults and children are underestimated by 30-50%. Animal protein production is "more resource intensive than any other form of food production" and their high saturated fat content is linked to chronic diseases in developed nations. Plant protein sources are important alternatives shown to "enhance ecosystem resilience and improve human health". Maize, commonly known as corn, is a staple food in the diets of more than 300 million Africans and ranks as the third most produced food globally. Maize supplies up to 80% of daily energy in sub-Saharan and Southern Africa alone. It is one of the main protein sources in these countries for vegetarians. Already, over 900,000 Canadians adults are vegetarians and globally plant protein consumption is encouraged. However, maize protein is limiting in the essential amino acid (EAA) tryptophan and anti-nutritional factors can affect tryptophan bioavailability (BA). Dietary protein quality (DPQ) depends on its amino acid (AA) composition and BA. Therefore, knowledge of tryptophan BA is fundamental to understand the extent to which cereal grains meet the body's requirement for protein synthesis (PS). Efforts aimed at increasing crop production and DPQ, should coincide with DPQ evaluation directly in humans so that the gap in knowledge between protein requirement and how best to provide it can be quickly and efficiently reconciled.

DETAILED DESCRIPTION:
Protein quality evaluation assesses the capacity of food proteins to meet the EAA needs of the body. The DPQ of plant proteins have been little studied in humans despite their importance in the diet and their well-recognized positive effects on chronic diseases. Dietary guidelines are encouraging increased plant protein consumption due to the benefits of plant protein. With the increasing interest in vegetarian diets in North America, it is imperative that the DPQ of cereal grains be evaluated so that plant protein recommendations are accompanied by an empirical understanding of plant protein quality. The information gathered from this project will provide additional experimental data in humans on plant protein quality (have completed lentils and chickpeas), on which nutrition recommendations can be built. Globally, this will also help support the FAO's commitment to compile tables on AABA of foods for global distribution. The aim of the study is to apply the IAAO method to determine the MA of tryptophan in maize prepared by moist cooking method.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 to 90 years old.
* In good general health as evidenced by medical history, physical health and blood draw.
* Fasting blood glucose, hemoglobin A1c (HbA1c), urea, creatinine.
* Willingness to participate in the study.
* BMI <30 kg/m2.

Exclusion Criteria:

* Presence of chronic disease and/or acute illness known to affect protein/amino acid metabolism (e.g. HIV, diabetes, taking medications known to affect protein/AA metabolism (e.g. steroids).

  * Inability to tolerate the diet (i.e. allergy).
  * Significant weight loss during the past month or consumption of weight reducing diets.
  * Significant caffeine consumption (>2 cups per day).
  * Significant consumption of alcohol (>1 drink per day i.e. 1 beer or ½ glass of wine).
  * Unwilling to have blood drawn from a venous access or using a ventilated hood indirect calorimeter for the purposes of the study.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-29 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-02 (Estimated)

PRIMARY OUTCOMES:
MA of tryptophan in maize | Up to 24 months
  To measure the tryptophan metabolic availability investigators will collect breath samples from participants. From these samples, investigators will measure the amount of amino acids oxidized and how much is retained in the body when graded intakes of tryptophan are consumed by the participants consuming a controlled diet.

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Courtney Martin, PhD, RD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No